CLINICAL TRIAL: NCT00370019
Title: Effect of Transdermal Estradiol Replacement Therapy on Ovulation Rate in Women With Premature Ovarian Failure: A Randomized, Placebo-Controlled Trial
Brief Title: Effects of an Estrogen Replacement Therapy Skin Patch on Ovulation in Women With Premature Ovarian Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Lawrence M. Nelson, M.D./National Institute of Child Health and Human Development, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060201; 06-CH-0201
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-12

CONDITIONS: Premature Ovarian Failure
Keywords: Premature Ovarian Failure; Ovulation; Fertility; Estrogen Replacement; Follicle Function; Premature Menopause; POF
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature | interventions — Lunelle

INTERVENTIONS:
Drug: Estradiol/Medroxyprogesterone acetate

SUMMARY:
This study will determine whether giving estrogen replacement therapy through an estradiol patch can improve ovulation rates in women with spontaneous premature ovarian failure. The ovaries are glands in women that produce female hormones and normally release an egg once a month. In women with spontaneous premature ovarian failure, the ovaries stop working too soon. Women with this disorder have abnormally high levels of leuteinizing hormone (LH) in their blood, which impedes normal ovulation. In some women, estrogen replacement can suppress LH levels to the normal range.

Women between 18 and 40 years of age with premature ovarian failure may be eligible for this 4-month study. Participants receive either standard hormone replacement therapy, consisting of an estradiol patch and progestin tablets, or placebo. The placebo group receives patches and tablets that look the same as those for the group with active treatment but they contain no hormone. All participants wear the patch every day and take the tablets the first 12 days of each month. In addition to taking the study drug, participants have blood drawn once a week for the 16 weeks of the study.

At the end of the trial, women who were in the placebo group are offered the opportunity to receive the estrogen patch and progestin therapy for another 16 weeks and continue the blood tests to determine if they ovulate on this treatment.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) is a life altering and distressing diagnosis for women due to associated infertility. Despite having amenorrhea and markedly elevated serum gonadotropin levels, approximately 50% of women with 46XX spontaneous premature ovarian failure have ovarian follicles that function intermittently. These follicles are faced with high serum LH levels. Normally, women have their LH levels in the range of 3-14 u/L except in the preovulatory stage, when it rises above 20 u/L. At that level it works on LH receptors on the granulosa cells and transforms the follicle in the corpus leutium. In POF, continuous high level of LH prematurely lutienizes growing follicles and thereby causes follicle dysfunction. We have shown by histological examination that inappropriate luteinization is a major mechanism of Graffian follicle dysfunction in these women.

We have found that approximately 50% women with premature ovarian failure have LH levels in the normal range while they are taking 100 mcg per day of our standardized transdermal estradiol therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with karyotypically normal spontaneous premature ovarian failure (as defined by screening protocol 91-CH-0127), i.e. women who have at least 4 months of amenorrhea, two FSH levels above 40 mIU/mL, or in the menopausal range, at least one month apart, and a normal 46, XX karyotype, diagnosed with premature ovarian failure prior to the age of 40 who are between the age of 18 and 40 years will be candidates.

Patients will be screened under the protocol 91-CH-0127 (Ovarian follicle function in patients with karyotypically normal spontaneous premature ovarian failure).

EXCLUSION CRITERIA:

1. General smokers (greater than 2 cigarettes/d), alcohol users (greater than 2 drinks/d), body mass index (BMI, kg/m(2) greater than or equal to 30 and less than or equal to 19, major dermatologic disorders, or a history of skin sensitivity to adhesive bandages, tape or transdermal matrix patches
2. Hysterectomy
3. Medication use current and/or past use of: diuretics, anticoagulants (heparin, coumadin), glucocorticoid drugs, gonadotropin-releasing hormone agonist or antagonist therapy, chemotherapy, use of other therapies to induce ovulation such as clomiphene citrate and other assisted reproductive technologies.(At present there are no proven ways to improve ovulation rate in these women)
4. Medical history of anorexia nervosa, hyperprolactinemia, Cushing's syndrome, gastrectomy, osteogenesis imperfecta, mastocytosis, rheumatoid arthritis, long term parenteral nutrition, hemolytic anemia, hemochromatosis and thalassemia, ankylosing spondylitis, multiple myeloma, any cancer, any other major illness
5. Contraindications to hormone replacement therapy thromboembolic event associated with previous estrogen use history of endometrial cancer or hyperplasia history of breast cancer

hypertriglyceridemia (fasting triglyceride levels greater than 250 mg/dL) undiagnosed vaginal bleeding known sensitivity to agents.

Active liver disease with more than 3 times elevation of liver enzymes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08-25; Primary Completion 2011-12-12 (Actual); Study Completion 2011-12-12 (Actual)

PRIMARY OUTCOMES:
Serum progesterone in the ovulatory range.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kreiner D, Droesch K, Navot D, Scott R, Rosenwaks Z. Spontaneous and pharmacologically induced remissions in patients with premature ovarian failure. Obstet Gynecol. 1988 Dec;72(6):926-8. doi: 10.1097/00006250-198812000-00024. PMID 3141855
- [Background] Santoro N, Schmidt CL. Pregnancy after an unsuccessful oocyte donation cycle. Fertil Steril. 1990 Jan;53(1):174-6. doi: 10.1016/s0015-0282(16)53238-5. PMID 2295340
- [Background] Wright CS, Jacobs HS. Spontaneous pregnancy in a patient with hypergonadotrophic ovarian failure. Br J Obstet Gynaecol. 1979 May;86(5):389-92. doi: 10.1111/j.1471-0528.1979.tb10617.x. PMID 556232